CLINICAL TRIAL: NCT05255094
Title: A Phase 3 Clinical Study Evaluating the Efficacy and Safety of AK102 in Patients With Primary Hypercholesterolemia and Mixed Hyperlipidemia
Brief Title: A Study to Evaluate the Efficacy and Safety of AK102 in Patients With Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK102-301
Record Dates: First submitted 2022-02-09; First posted 2022-02-24 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AK102 regimen 1 (Experimental)
  Interventions: Biological: AK102
- AK102 regimen 2 (Experimental)
  Interventions: Biological: AK102
- Placebo 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AK102 — Administered AK102 by subcutaneous injection every 2 weeks Drug: Statins and/or Ezetimibe lipid-lowering therapies
  Arms: AK102 regimen 1
Biological: AK102 — Administered AK102 by subcutaneous injection every 4 weeks Drug: Statins and/or Ezetimibe lipid-lowering therapies
  Arms: AK102 regimen 2
Drug: Placebo — Administered placebo by subcutaneous injection every 2 weeks Drug: Statins and/or Ezetimibe lipid-lowering therapies
  Arms: Placebo 1
Drug: Placebo — Administered placebo by subcutaneous injection every 4 weeks Drug: Statins and/or Ezetimibe lipid-lowering therapies
  Arms: Placebo 2

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 3 clinical study evaluating the efficacy and safety of AK102 in patients with primary hypercholesterolemia and mixed hyperlipidemia.

DETAILED DESCRIPTION:
This is a Phase 3 clinical study to evaluate the efficacy and safety of AK102, a monoclonal antibody against proprotein convertase subtilisin/kexin type 9 (PCSK9), in subjects with primary hypercholesterolemia and mixed hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject understand and voluntarily sign the written Inform Consent Form (ICF).
2. Male or female ≥ 18 to ≤ 80 years of age.
3. The fasting serum LDL-C level of subjects did not meet the treatment goal after at least 4 weeks of stable lipid-lowering background treatment.
4. TG ≤ 4.5 mmol/L (400 mg/dl).

Exclusion Criteria:

1. Known homozygous familial hypercholesterolemia.
2. Received PCSK9 inhibitors within 6 months before randomization.
3. Known sensitivity to PCSK9 inhibitors and any substances to be administered.
4. Severe renal dysfunction.
5. Previously received organ transplantation.
6. Uncontrolled hypothyroidism or hyperthyroidism.
7. Uncontrolled hypertension.
8. Known hyperlipidemia secondary to comorbidity, including nephrotic syndrome, cholestatic liver failure, etc.
9. History of malignancy of any organ system within the past 5 years.
10. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline of serum LDL-C level | At week 12
  Percentage change from baseline of serum LDL-C level

SECONDARY OUTCOMES:
Percentage change from baseline of serum TC, HDL-C, TG, ApoB, ApoA-I, non HDL-C and Lp(a) levels | Week 0-12
  Percentage change from baseline of serum TC, HDL-C, TG, ApoB, ApoA-I, non HDL-
The incidence and severity of adverse events (AE) | Week 0-12
  The incidence and severity of adverse events (AE)
To evaluate the population pharmacokinetic (PK) characteristics of AK102，such as AK102 concentration | Week 0-12
  To evaluate the population pharmacokinetic (PK) characteristics of AK102，such as AK102 concentration
Number and percentage of subjects with positive anti-ak102 antibody (ADA) / neutralizing antibody (NAB) and the time of ADA / nab positivity | Week 0-12
  Number and percentage of subjects with positive anti-ak102 antibody (ADA) / neutralizing antibody (NAB) and the time of ADA / nab positivity

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No